CLINICAL TRIAL: NCT03735134
Title: Colchicine in Periprocedural Myocardial Infarction: the Role of Alpha Defensin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HYMC-99-18
Record Dates: First submitted 2018-11-07; First posted 2018-11-08 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Inflammation; Myocardial Infarction
MeSH Terms: conditions — Inflammation; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Active Comparator): Stable coronary artery disease patients who have been assigned to elective PCI and who will be given standard of care treatment
  Interventions: Drug: Standard of care treatment prior to elective PCI
- Early colchicine loading dose (Active Comparator): Stable coronary artery disease patients who have been assigned to elective PCI and who will be given standard of care treatment plus colchicine loading dose 12-24 hours before PCI
  Interventions: Drug: Colchicine Loading Dose
- Late colchicine loading dose (Active Comparator): Stable coronary artery disease patients who have been assigned to elective PCI and who will be given standard of care treatment plus colchicine loading dose one hour prior to PCI
  Interventions: Drug: Colchicine Loading Dose

INTERVENTIONS:
Drug: Colchicine Loading Dose — Two milligrams of colchicine will be administrated in addition to the standard of care treatment
  Arms: Early colchicine loading dose; Late colchicine loading dose
Drug: Standard of care treatment prior to elective PCI — All medications normally given to patients prior to elective PCI
  Arms: Control Group

SUMMARY:
The aim of this research is to study the effect of a loading dose of colchicine on the occurrence of periprocedural myocardial infarction (PPMI) in elective percutaneous coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized with troponin negative events and scheduled for elective PCI

Exclusion Criteria:

* Significant renal dysfunction
* Significant liver dysfunction
* Severe left ventricular dysfunction
* Severe low weight
* Chronic colchicine treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Occurrence of PPMI post elective PCI | 24 hours post PCI
  Occurrence of PPMI post elective PCI and its relation to defensin levels

SECONDARY OUTCOMES:
Traditional inflammatory markers | 24 hours post PCI
  Determination of traditional inflammatory markers including c-reactive protein, white blood cells and interleukin-6
Major adverse cardiovascular events | 30 days
  Determining the occurrence of major adverse cardiovascular events

CONTACTS AND LOCATIONS:
Locations (1):
- Hille Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No